CLINICAL TRIAL: NCT05605067
Title: Genetic Architecture of Avoidant/Restrictive Food Intake Disorder
Acronym: ARFID-GEN
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Psychiatric Center Ballerup (Other)
Responsible Party: Sponsor
Other Study IDs: 22-1524; R56MH129437 (NIH)
Record Dates: First submitted 2022-10-26; First posted 2022-11-04 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-08

CONDITIONS: ARFID; Eating Disorders; Eating Disorders in Children; Eating, Picky
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Feeding and Eating Disorders; Food Fussiness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples from participants for DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Participants will self-select into the study. All enrolled will meet study specific criteria and be considered cases.

SUMMARY:
The goal of this observational study is to rapidly accelerate knowledge about the biology of avoidant and restrictive food intake disorder or ARFID in children ages 7-17 and in adults. The investigators will be evaluating the genetic and environmental origins of ARFID. Participants will be asked to answer questionnaires online and to submit a saliva sample for DNA using a kit that will be mailed to their home.

ELIGIBILITY:
Inclusion Criteria:

* Meet study criteria for ARFID
* Be willing to submit a saliva sample
* Have a US mailing address
* English-speaking

Exclusion Criteria:

* Potential other eating disorders

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents of children with ARFID and adults with ARFID will self-select into the study. Because the study is conducted online, participants can join from across the United States
Sampling Method: Non-Probability Sample
Enrollment: 5076 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Case definitions | Baseline
  Number of enrolled individuals who meet the case definition

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Bulik, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The specimens (saliva and DNA) and data (from questionnaires) may be shared with researchers at UNC or other institutions, such as the National Institutes of Health (NIH), and will eventually be included in the NIH data repository without additional consent. Research studies may be done at many places at the same time. No personal, identifying information will be sent to other researchers or included in the data repository. To secure the data, the NIH data repository will include multiple tiers of data security such as sequential firewalls, independent networks, and encryption based on the content and level of risk associated with the data. All data and information will be submitted to a high security network within NIH through a secure transmission process.
  No participant will be identified in any report or publication about research using their specimens.
Supporting Information: ICF
Time Frame: Questionnaire data and saliva samples will be submitted to NIMH repositories within 6 months after end of study. Genetic results will be submitted within one year after initial publication. All data will be available after the respective embargo periods.
Access Criteria: https://dbgap.ncbi.nlm.nih.gov/aa/dbgap_request_process.pdf https://nda.nih.gov/nda/access-data-info.html

REFERENCES:
- [Derived] Bulik CM, Micali N, MacDermod CM, Qi B, Munn-Chernoff MA, Thornton LM, White J, Dinkler L, Pisetsky EM, Johnson J, Devine KR, Ortiz SN, Silverman AE, Berthold N, Dumain A, Guintivano J, Halvorsen M, Crowley JJ. ARFID Genes and Environment (ARFID-GEN): study protocol. BMC Psychiatry. 2023 Nov 21;23(1):863. doi: 10.1186/s12888-023-05266-x. PMID 37990202
- [Derived] Bulik CM, Micali N, MacDermod CM, Qi B, Munn-Chernoff MA, Thornton LM, White J, Dinkler L, Pisetsky EM, Johnson J, Devine KR, Ortiz SN, Silverman AE, Berthold N, Dumain A, Guintivano J, Halvorsen M, James J. Arfid Genes and Environment (ARFID-GEN): Study Protocol. Res Sq [Preprint]. 2023 Aug 31:rs.3.rs-3186174. doi: 10.21203/rs.3.rs-3186174/v1. PMID 37693386